CLINICAL TRIAL: NCT03128567
Title: Effets de la Stimulation cérébrale Profonde Chez Les Patients âgés Avec Maladie de Parkinson : Essai contrôlé randomisé Multicentrique
Brief Title: Deep Brain Stimulation for Patients With Parkinson's Disease.
Acronym: STTARTLATE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C 14-01
Record Dates: First submitted 2017-02-23; First posted 2017-04-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stimulation of the subthalamic nucleus: 25 patients with Parkinson's disease
  Interventions: Device: Stimulation of the subthalamic nucleus
- Best medical treatment: 25 patients with Parkinson's disease

INTERVENTIONS:
Device: Stimulation of the subthalamic nucleus — Stimulation of the subthalamic nucleus
  Groups: Stimulation of the subthalamic nucleus

SUMMARY:
Deep brain stimulation of the sub thalamic nucleus (STN-DBS) is an efficient treatment to improve motor and non motor signs of Parkinson's disease (PD). In people aged more 70 years, an increased rate of side effects such as post-operative cognitive decline and/or postural instability with falls has been suspected with less improvement in the quality of life. Here, Investigators aim further explore the effects of STN-DBS in 50 patients with PD people aged more 69 years in a randomized parallel controlled study.

DETAILED DESCRIPTION:
The effects of combined bilateral deep brain stimulation of the subthalamic nucleus and medical treatment on the quality of life will be evaluated in 25 PD patients aged more 69 years in comparison to 25 PD patients aged more 69 years that only received medical drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* disease duration > 5 years
* levodopa related motor complications
* dopasensitivity > 50%
* signed informed written consent
* medical social insurance

Exclusion Criteria:

* dementia
* contra-indication to neurosurgery

Ages: 69 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
PDQ-39 Quality of life questionnary | Quality of life one year after surgery
  PDQ-39 scale

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service d'EFSN, Hôpital Pellegrin, Bordeaux
  - Hôpital Roger Salengro - CHRU de Lille Service de Neurologie et Pathologie du Mouvement, Lille
  - Hôpital Neurologique Pierre Wertheimer, Service de Neurologie, Lyon
  - Département des maladies du Système Nerveux, Hôpital Pitié-Salpétrière, Paris
  - Service de Neurologie, Pôle Neurosciences, CHU de Poitiers, Poitiers
  - CHU Charles Nicolle, Rouen
  - Centre d'Investigation Clinique - CIC 1436. CHU PURPAN. Hôpital Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No